

Title: Specified Drug-Use Survey ("Long-Term Use Survey") on Zacras Combination

Tablets LD & HD

NCT Number: NCT02181816

Protocol Approve Date: 02-Jun-2017

Certain information within this protocol has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally

identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

Named persons or organizations associated with the study.

Patient identifiers within the text, tables, or figures or in by-patient data listings.

Proprietary information, such as scales or coding systems, which are considered

confidential information under prior agreements with license holder.

Other information as needed to protect confidentiality of Takeda or partners,

personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable

information or company confidential information may be removed in their entirety if it

is considered that they do not add substantially to the interpretation of the data (eg,

appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version

was Japanese.

## Protocol for Specified Drug-Use Survey Specified Drug-Use Survey ("Long-Term Use Survey") on Zacras Combination Tablets LD & HD

Version number 4th version
Date of 2 June 2017

preparation

**Sponsor** Takeda Pharmaceutical Company Limited

#### Table of Contents

| 1.0 | | Bacl | kground | 4 |
|---|---|---|---|---|
| 2.0 | | Obje | ectives | 2 |
| 3.0 | | Plan | ned Sample Size and Rationale | 2 |
| 3.1 | 1 | Plan | ned Sample Size | 2 |
| 3.2 | 2 | Rati | onale | 2 |
| 4.0 | | Surv | rey Population | 4 |
| 4.1 | 1 | Excl | usion Criteria | 4 |
| 5.0 | | Dosa | age and Administration | 4 |
| 6.0 | | Plan | ned Number of Medical Institutions by Department | ( |
| 7.0 | | Met | hods | ( |
| 7.1 | 1 | Obs | ervation Period | ( |
| 7.2 | 2 | Req | uest to and Contract with the Study Site | ( |
| 7.3 | 3 | Met | hod of Patient Registration | ( |
| 7.4 | 4 | Con | pletion and Submission of Case Report Form | |
| 7.5 | 5 | Acti | ons to be Taken in Case of Serious Adverse Events | 7 |
| 8.0 | | Plan | ned Period | |
| 9.0 | | Surv | vey Items | |
| 9.1 | 1 | Entr | ies into the Patient Registration Form | |
| 9.2 | 2 | Entr | ies into the Case Report Form | 8 |
| | 9.2.1 | 1 Cover of the Case Report Form | | |
| | 9.2.2 | 2 | Patient Demographics and Baseline Characteristics | 8 |
| 9.2.2<br>9.2.3 | | 3 Treatment Given | | |
| | 9.2.4 | ļ | Tests/Observations | 8 |
| | 9.2.4 | 1.1 | Vital Signs | 8 |
| | 9.2.4 | 1.2 | Laboratory Tests | 9 |
| | 9.2.4 | 1.3 | Other Observations | 9 |
| | 9.2.5 | 5 | Adverse Events (AEs) | 9 |
| 10.0 | | Ana | lysis Items and Methods | 11 |
| 10 | 1.1 | Matt | ters on Patient Composition1 | 11 |
| 10 | .2 | Patie | ent Demographics and Baseline Characteristics | 11 |
| 10 | | | tment Given1 | |
| 10 | .4 | Mat | ters on Safety | 1 |
| | 10.4 | .1 | Occurrence of Adverse Events | . 2 |
| | 10.4 | .2 | Factors that May Affect the Safety | . 2 |
| 10 | .5 | | ters on Efficacy | |
| | 10.5 | | Office Blood Pressure | |
| | 10.5 | .2 | Factors that May Affect the Efficacy | |
| 11.0 | | Post | ing of Survey Information | |
| 12.0 | | | anization 1 | , |

| 12.1 | Administrative Manager | 12 |
|----------|------------------------------------------------|----|
| 12.2 | Central Registration Center | 12 |
| 13.0 | Contract Research Organization | 13 |
| 14.0 | Other Necessary Matters | 13 |
| 14.1 | Revision of the Protocol | 13 |
| 14.2 | Actions to be Taken for Problems and Questions | 13 |
| Appendix | x Observation schedule | |

#### 1.0 Background

Since drugs for hypertension are generally used for a long period of time, the safety of long-term use must be established. While the safety of long-term use of Zacras Combination Tablets LD & HD (hereinafter referred to as Zacras Combination Tablets) was already evaluated in a Japanese Phase III long-term clinical study (duration of treatment: 52 weeks, number of evaluated subjects: 368), it is necessary to evaluate the safety in more patients in clinical settings after marketing, a population that, unlike the study population, receive the drug in diverse situations.

Accordingly, a specified drug-use survey (hereinafter referred to as the survey) is planned to evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in hypertensive patients in daily medical practice. This survey will be conducted in compliance with Good Post-marketing Study Practice (GPSP) ordinance and related requirements.

#### 2.0 Objectives

To evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in hypertensive patients in daily medical practice

#### 3.0 Planned Sample Size and Rationale

#### 3.1 Planned Sample Size

1,000 patients

#### 3.2 Rationale

Patient populations identified as important missing information from Japanese clinical studies of Zacras Combination Tablets are patients with renal impairment, patients with hepatic impairment, and elderly patients ( $\geq 75$  years old). The sample size required to evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in these patient populations was calculated by reference to previous results. More specifically, according to final tabulation (number of patients included in safety evaluation: 3,300) in a previous specified drug-use survey (long-term use survey in hypertension) of a fixed-dose combination (UNISIA Combination Tablets) of an angiotensin receptor blocker (ARB) (candesartan) and a Ca antagonist (amlodipine), which belongs to the pharmacologically same class as Zacras Combination Tablets, patients with renal impairment, patients with hepatic impairment, and elderly patients (and those  $\geq$ 75 years old) accounted for 6.9%, 11.5%, and 65.2% (36.8%) of all patients, respectively. According to final tabulation (number of patients included in safety evaluation: 4,152) in a drug use-results survey of candesartan alone (BLOPRESS Tablets), patients with renal impairment, patients with hepatic impairment, and elderly patients (and those  $\geq 75$  years old) accounted for 9.5%, 10.6%, and 53.2% (22.1%), respectively. With a target sample size of 1,000 patients for the present survey, 70 patients with renal impairment, 100 patients with hepatic impairment, and 500 elderly patients (and 200 patients ≥75 years old)

are expected to be collected, probably allowing the safety and efficacy evaluation in these populations. This calculation is not based on statistical estimation.

#### 4.0 Survey Population

The survey population consists of hypertensive patients who do not meet any of the exclusion criteria listed in Section 4.1. Refer to the "Precautions for Indication" (presented below) and "Precautions" sections in the package insert.

<Pre><Precautions for Indication>

Zacras Combination Tablets should not be used as the first-line treatment of hypertension. An excessive drop in blood pressure may occur.

#### 4.1 Exclusion Criteria

Patients who meet any of the following criteria should be excluded from the survey:

- (1) Patients with a history of hypersensitivity to any of the ingredients of Zacras Combination Tablets or other dihydropyridines
- (2) Patients who are or may be pregnant
- (3) Diabetic patients taking aliskiren fumarate (excluding those with markedly poor blood pressure control despite other antihypertensive treatments)

#### 5.0 Dosage and Administration

For adults, one Zacras Combination Tablet (20 mg/2.5 mg or 20 mg/5 mg of azilsartan/amlodipine) will be administered orally once daily. Zacras Combination Tablets should not be used as the first-line treatment of hypertension. Refer to the "Precautions for Dosage and Administration" (presented below) and "Precautions" sections in the package insert.

<Precautions for Dosage and Administration>

(1) It should be determined whether Zacras Combination Tablets are indicated for each patient individually based on the following Dosage and Administration and Precautions for Dosage and Administration of azilsartan and amlodipine besilate, as well as other relevant information:

Azilsartan

Dosage and Administration

For adults, azilsartan 20 mg should usually be administered orally once daily. The dose may be increased or reduced as appropriate based on age and symptoms, with the maximum daily dose being 40 mg.

Precautions for Dosage and Administration

It should be carefully determined whether or not azilsartan is indicated while keeping the hypotensive effect of azilsartan in mind. Initiation of treatment at a low dose below 20 mg should also be considered.

Amlodipine besilate

•Hypertension

Dosage and Administration

For adults, amlodipine 2.5 to 5 mg should usually be administered orally once daily. The dose may be increased or reduced as appropriate based on symptoms. In the case of insufficient response, the dose may be increased up to 10 mg given once daily.

- (2) As a general rule, switching to Zacras Combination Tablets should be considered for patients receiving azilsartan 20 mg with amlodipine 2.5 to 5 mg or patients with poor blood pressure control despite treatment with either one of these treatments.
- 6.0 Planned Number of Medical Institutions by Department

Internal medicine and other departments Approximately 250 medical institutions

- 7.0 Methods
  - 7.1 Observation Period

12 months

#### 7.2 Request to and Contract with the Study Site

Request and contract for participation in the survey will be made using a paper case report form (CRF). A representative of Takeda Pharmaceutical Company Limited (hereinafter referred to as Takeda's representative) will explain the objectives, contents, and methods of the survey to the investigator based on "Request for cooperation for specified drug-use survey," "Implementation outline," "Patient registration form (sample)," and "Case report form (sample)" to enter into a written contract with the study site and request the study site to conduct a survey within a specified period.

#### 7.3 Method of Patient Registration

Patients will be registered using the central registration system via fax. After the start of the contract with the study site, the investigator shall register each patient for whom Zacras Combination Tablets are prescribed by faxing a patient registration form containing patient registration information (refer to Section 9.1) to the central registration center (refer to Section 12.2) within 14 days after prescription of Zacras Combination Tablets (day of prescription designated as day 0 and day following the day of prescription designated as 1 day after prescription). No patient can be registered before Zacras Combination Tablets are actually prescribed. Patients determined by the central registration center to be ineligible for any reason cannot be registered. The investigator shall register a new patient using a new patient registration form supplied by Takeda's representative.

Takeda's representative will supply a CRF, which will be issued after the central registration

center decides to register the relevant patient, to the investigator.

#### 7.4 Completion and Submission of Case Report Form

For each of all registered patients, the investigator shall complete and submit a CRF to Takeda Pharmaceutical within approximately 1 month after the end of the observation period. Any failure to confirm the intake of Zacras Combination Tablets shall be specified (no further information is required).

For patients discontinued from treatment with Zacras Combination Tablets for any reason during the observation period, the investigator shall complete and submit a CRF to Takeda Pharmaceutical within approximately 1 month after the end of required observation. For any patient discontinued from treatment with Zacras Combination Tablets due to an adverse event, the investigator shall complete and submit a CRF to Takeda Pharmaceutical after monitoring the patient as long after discontinuation of treatment as possible until the adverse event is confirmed to have resolved or be resolving.

#### 7.5 Actions to be Taken in Case of Serious Adverse Events

The investigator shall immediately communicate any serious adverse event in the observation period to Takeda's representative. In addition, the investigator shall provide detailed information at the request of Takeda's representative.

#### 8.0 Planned Period

Survey period: From June 2014 to 31 January 2017

Patient enrollment period: From June 2014 to 31 January 2016<sup>Note)</sup>

Note) Patient registration (receipt of a patient registration form via fax) will not be accepted on 1 February 2016 onwards even if Zacras Combination Tablets are prescribed by 31 January 2016.

If the number of patients enrolled in the survey reaches the planned sample size before 31 January 2016, acceptance of registration will be terminated before the end of the patient enrollment period. If the patient enrollment period is shortened, the survey period will be changed accordingly.

#### 9.0 Survey Items

The investigator shall enter the items listed below into the patient registration form and the CRF. The survey schedule is presented in Appendix.

#### 9.1 Entries into the Patient Registration Form

#### 1) Survey items

Name of the medical institution, name of a physician who completes the patient registration form, date of prescription of Zacras Combination Tablets, patient identification number, patient initials, sex, date of birth, assessment based on the inclusion criteria, assessment

based on the exclusion criteria, presence or absence of breast-feeding (only females)

2) Time points of survey

At patient registration

#### 9.2 Entries into the Case Report Form

#### 9.2.1 Cover of the Case Report Form

Date of final entry into the CRF, name of a physician who completes the CRF

#### 9.2.2 Patient Demographics and Baseline Characteristics

#### 1) Survey items

Time of diagnosis of hypertension, diagnostic category (at the start of treatment with Zacras Combination Tablets), predisposition to hypersensitivity (presence or absence and details), concurrent illness (presence or absence and details), medical history (presence or absence and details), height, body weight, smoking history, drinking history, presence or absence of breast-feeding (at the start of treatment with Zacras Combination Tablets) [only females]

2) Time points of survey

At the start of treatment with Zacras Combination Tablets

#### 9.2.3 Treatment Given

#### 1) Survey items

Details on the use of Zacras Combination Tablets (daily dose, duration of treatment, and reason for discontinuation of treatment), details on the use of other antihypertensive \* (presence or absence, name of the drug, daily dose, and duration of treatment), details on the use of concomitant non-antihypertensive drug (presence or absence, name of the drug, and purpose of use)

#### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

\* Period from 2 months before the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment) for details on the use of other antihypertensive

#### 9.2.4 Tests/Observations

#### 9.2.4.1 Vital Signs

1) Tests/observations

Office blood pressure (systolic/diastolic), pulse rate

2) Time points of survey

Time points of measurement at the start of treatment with Zacras Combination Tablets and after 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 months of treatment (or discontinuation of

treatment)

#### 9.2.4.2 Laboratory Tests

#### 1) Test parameters

White blood cell count, platelet count, aspartate aminotransferase (AST), alanine aminotransferase (ALT),  $\gamma$ -glutamyl transpeptidase ( $\gamma$ -GTP), serum creatinine, blood urea nitrogen (BUN), serum potassium

#### 2) Time points of survey

Time points of test from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

#### 9.2.4.3 Other Observations

#### 1) Observations

Presence or absence of pregnancy in the observation period (only females)

If pregnancy is detected during the observation period, treatment with Zacras Combination

Tablets should be discontinued immediately, and Takeda's representative should be

informed. The investigator shall provide detailed information (including information up to
delivery such as premature delivery, wherever possible) using a pregnancy sheet at the
request of Takeda's representative.

#### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

#### 9.2.5 Adverse Events (AEs)

#### 1) Survey items

Presence or absence of AE (refer to Table 1), AE term, date of onset, seriousness and reason for seriousness (refer to Table 2), presence or absence of discontinuation of treatment with Zacras Combination Tablets, date of outcome assessment, outcome, causal relationship to Zacras Combination Tablets\* (refer to Table 3)

Patients with "not resolved" or "unknown" outcome or "unevaluable" causal relationship should be followed up wherever possible.

#### Note) Additional points to consider for AEs

Abnormal worsening of target disease, for instance, worsening beyond the expected natural course of the disease, will be handled as an AE, but expected worsening of target disease should not be handled as an AE.

#### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of

<sup>\*</sup> For the causal relationship to Zacras Combination Tablets, the rationale for "not related" and the reason for "unevaluable" shall be collected.

#### Table 1 Definition of adverse events

An AE is defined as any untoward medical occurrence in a clinical investigation subject administered a drug; it does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavorable or unintended sign (e.g., abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.

The following are also handled as AEs:

- •Symptoms and so forth that occur in infants breast-fed by their mothers under treatment with a drug
- •Symptoms and so forth that occur in children treated with a drug
- · Symptoms and so forth that occur as a result of occupational exposure to a drug
- · Symptoms and so forth that occur after administration of counterfeit medicines of our ethical drugs

#### Table 2 Criteria for assessing seriousness

An AE satisfying any of the following is assessed as serious:

- 1. Results in death (death)
- 2. Is life-threatening (risk of death)
- 3. Requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization/prolonged hospitalization)
- 4. Results in persistent or significant disability/incapacity (disability)
- 5. Leads to a congenital anomaly/birth defect (congenital anomaly)
- 6. Is an important medical event according to 1 to 5 described above, including AEs in Takeda Medically Significant AE List

#### Takeda Medically Significant AE List

Acute liver failure

| Takeda Medically Significant AE List | |
|---|---|
| •Acute respiratory failure/acute respiratory distress | •Anaphylactic shock |
| syndrome (ARDS) | |
| •Torsade de pointes / ventricular fibrillation / ventricular | •Acute renal failure |
| tachycardia | |
| •Malignant hypertension | •Pulmonary hypertension |
| •Convulsive seizures (including convulsion and epilepsy) | •Pulmonary fibrosis (including interstitial |
| | pneumonia) |
| •Agranulocytosis | •Neuroleptic malignant syndrome / |
| | malignant hyperthermia |
| •Aplastic anemia | •Spontaneous abortion / stillbirth and fetal |
| | death |
| •Toxic epidermal necrolysis / oculomucocutaneous | •Confirmed or suspected transmission of |
| syndrome (Stevens-Johnson syndrome) | infectious agent by a medicinal product |
| •Hepatic necrosis | •Confirmed or suspected endotoxin shock |

Table 3 Criteria for assessing the relationship of each adverse event to Zacras Combination Tablets

| Assessment | Criteria for assessment |
|---|---|
| | An AE that follows a reasonable temporal sequence from |
| | administration of a drug (including the course after withdrawal of the |
| Dalata d | drug), or for which possible involvement of the drug can be argued, |
| Related | although factors other than the drug, such as underlying diseases, |
| | concurrent illnesses, concomitant drugs, and concomitant treatments, |
| | may also be responsible |
| | An AE that does not follow a reasonable temporal sequence from |
| | administration of a drug and/or that can reasonably be explained by |
| Not related | other factors, such as underlying diseases, concurrent illnesses, |
| | concomitant drugs, and concomitant treatments |
| | Information necessary for evaluation, including temporal sequence |
| T. 1 11 | from administration of a drug (including the course after withdrawal |
| Unevaluable | of the drug), underlying diseases, concurrent illnesses, concomitant |
| | drugs, and concomitant treatments, is not sufficient. |

#### 10.0 Analysis Items and Methods

#### 10.1 Matters on Patient Composition

The number of enrolled patients, number of patients from whom the CRF is collected, number of patients included in safety/efficacy analysis, number of patients excluded from analysis, and reason for exclusion will be tabulated.

#### 10.2 Patient Demographics and Baseline Characteristics

Patient demographics and baseline characteristics, including sex, age, duration of disease, predisposition to hypersensitivity, and concurrent illness, will be tabulated.

#### 10.3 Treatment Given

Details on the use of Zacras Combination Tablets, details on the use of other antihypertensive, and details on the use of concomitant non-antihypertensive drug will be tabulated.

#### 10.4 Matters on Safety

For the safety analysis set, data will be tabulated as described below. AEs will be coded according to the MedDRA/J and summarized using preferred term (PT) and system organ class (SOC).

#### 10.4.1 Occurrence of Adverse Events

For AEs reported during the observation period, the incidence will be tabulated by type, time of onset, seriousness, and causal relationship to Zacras Combination Tablets.

#### 10.4.2 Factors that May Affect the Safety

For AEs reported during the observation period, the incidence will be tabulated by patient background factors (e.g., sex, age, presence or absence of concurrent renal impairment, presence or absence of concurrent hepatic impairment) and treatment given (e.g., details on the use of Zacras Combination Tablets, details on the use of concomitant drug).

#### 10.5 Matters on Efficacy

For the efficacy analysis set, data will be tabulated as described below.

#### 10.5.1 Office Blood Pressure

For office blood pressure, measured value, change (measured value at each post-baseline time point of measurement - measured value at the start of treatment with Zacras Combination Tablets), and percentage change [(measured value at each time point of measurement - measured value at the start of treatment with Zacras Combination Tablets)  $\div$  measured value at the start of treatment with Zacras Combination Tablets  $\times$  100] at each time point of test will be tabulated.

#### 10.5.2 Factors that May Affect the Efficacy

Office blood pressure will be tabulated by patient background factors (e.g., sex, age) and treatment given (e.g., details on the use of Zacras Combination Tablets, details on the use of other antihypertensive).

#### 11.0 Posting of Survey Information

Takeda Pharmaceutical Company Limited will post survey information on Clinical Trials.gov and an open website (JAPIC-CTI\*) before starting the survey.

#### 12.0 Organization

| 1 ^ - | 1 4 1 | | | 3 4 | r |
|--------------|-------|-------|---------|---------|---------|
| ı ' <i>)</i> | 1 1 | lmini | atratix | 70 1/ | lanager |
| 12. | | | SHAH | v 🗁 ıvı | anaye |

PPD

Takeda Pharmaceutical Company Limited

### 12.2 Central Registration Center PPD

<sup>\*</sup> Japan Pharmaceutical Information Center-Clinical Trials Information



#### 14.0 Other Necessary Matters

#### 14.1 Revision of the Protocol

During the survey, attention will be paid to comprehend the status of progression of the survey, presence or absence of unexpected adverse drug reactions (ADRs)/serious ADRs (based on precautions), presence or absence of increased incidence of certain ADRs, and appropriateness of survey items, and this protocol will be reviewed and revised if necessary. If partial change to dosage and administration or indications is approved during the survey, the necessity of revising the protocol will be discussed if necessary, and the protocol will be revised as needed.

#### 14.2 Actions to be Taken for Problems and Questions

If any safety or efficacy problem is detected, data will be carefully examined to discuss measures.

#### Appendix Observation schedule

| Time point of survey | | | | | | | O | bserv | ation | perio | od | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time point of survey | | | | | | | | | | | | | ب | ر. | ب | of |
| Survey item | | At patient registration | Start of treatment | After 1 month of treatment | After 2 months of treatment | After 3 months of treatment | After 4 months of treatment | After 5 months of treatment | After 6 months of treatment | After 7 months of treatment | After 8 months of treatment | After 9 months of treatment | After 10 months of treatment | After 11 months of treatment | After 12 months of treatment | At discontinuation c treatment |
| | Date of prescription of Zacras | 0 | | | | | | | | | | | | | | |
| | Combination Tablets | 0 | | | | | | | | | | | | | | |
| ion | Patient identification number | 0 | | | | | | | | | | | | | | |
| strat | Patient initials | 0 | | | | | | | | | | | | | | |
| regi | Sex | 0 | | | | | | | | | | | | | | |
| Patient registration | Date of birth | 0 | | | | | | | | | | | | | | |
| Pati | Inclusion/exclusion criteria | 0 | | | | | | | | | | | | | | |
| | Presence or absence of | 0 | | | | | | | | | | | | | | |
| | breast-feeding (only females) | | | | | | | | | | | | | | | |
| ics | Time of diagnosis of | | 0 | | | | | | | | | | | | | |
| demographics and baseline characteristics | hypertension | | | | | | | | | | | | | | | |
| narac | Diagnostic category | | 0 | | | | | | | | | | | | | |
| ne cl | Predisposition to hypersensitivity | | 0 | | | | | | | | | | | | | |
| aseli | Concurrent illness | | 0 | | | | | | | | | | | | | |
| and b | Medical history | | 0 | | | | | | | | | | | | | |
| hics | Height, body weight | | 0 | | | | | | | | | | | | | |
| grap | Smoking history | | 0 | | | | | | | | | | | | | |
| demo | Drinking history | | 0 | | | | | | | | | | | | | |
| Patient | Presence or absence of | | 0 | | | | | | | | | | | | | |
| Pat | breast-feeding (only females) | | | | | | | | | | | | | | | |
| c. | Details on the use of Zacras | | _ | | | | | | 0 | | | | | | | . 0 |
| n, et | Combination Tablets | | • | | | | | | | ············· | 0 | | | | | |
| Treatment given, etc. | Details on the use of other | | _ | | | | | | 0 | | | | | | | . 0 |
| ent | antihypertensive | | | | | | | | | | | | | | | |
| eatır | Details on the use of concomitant | | | | | | | | | | | | | | | |
| Tr | non-antihypertensive drug | | • | | | | | | 0 | | | | | | | 0 |
| tc. | Office blood pressure | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Tests/observations, etc. | Pulse rate | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| ation | White blood cell count | | • | | | | | | 0 | | | | | | <b></b> | 0 |
| Serv | Platelet count | • | • | | | | | | 0 | | | | | | <b></b> | 0 |
| ts/ob | AST | | • | | | | | | 0 | | | | | | <b></b> | 0 |
| Tes | ALT | | • | | | | | | 0 | | | | | | <b></b> | 0 |
| - | | L | 4 | | | | | | | | | | | | | لل |

| γ-GTP | <b>4</b> | 0 | <b>\</b> |
|---|---|---|---|
| Serum creatinine | | 0 | • 0 |
| BUN | <b>←</b> | o | • 0 |
| Serum potassium | <b>—</b> | o | <b>&gt;</b> 0 |
| Presence or absence of pregnancy (only females) | <b>-</b> | o — | • 0 |
| Adverse event | 4 | o | <b>&gt;</b> 0 |

o : Performed

← ∘ Performed throughout the period

## Protocol for Specified Drug-Use Survey Specified Drug-Use Survey ("Long-Term Use Survey") on Zacras Combination Tablets LD & HD

Version number 3rd version
Date of 1 April 2015

preparation

**Sponsor** Takeda Pharmaceutical Company Limited

#### Table of Contents

| 1.0 | Bac | ckground | 4 |
|------|------|-----------------------------------------------------|----|
| 2.0 | Ob | jectives | 4 |
| 3.0 | Pla | nned Sample Size and Rationale | 4 |
| 3.1 | Pla | nned Sample Size | 4 |
| 3.2 | Rat | tionale | 4 |
| 4.0 | Sur | rvey Population | 5 |
| 4.1 | Exc | clusion Criteria | 5 |
| 5.0 | Do | sage and Administration | 5 |
| 6.0 | Pla | nned Number of Medical Institutions by Department | 6 |
| 7.0 | Me | ethods | 6 |
| 7.1 | Ob | servation Period | 6 |
| 7.2 | Red | quest to and Contract with the Study Site | 6 |
| 7.3 | Me | ethod of Patient Registration | 6 |
| 7.4 | Co | mpletion and Submission of Case Report Form | 7 |
| 7.5 | Act | tions to be Taken in Case of Serious Adverse Events | 7 |
| 8.0 | Pla | nned Period | 7 |
| 9.0 | Sur | rvey Items | 7 |
| 9.1 | Ent | tries into the Patient Registration Form | 7 |
| 9.2 | Ent | tries into the Case Report Form | 8 |
| 9.2 | 1 | Cover of the Case Report Form. | 8 |
| 9.2 | 2 | Patient Demographics and Baseline Characteristics | 8 |
| 9.2 | 3 | Treatment Given | 8 |
| 9.2 | .4 | Tests/Observations | 8 |
| 9.2 | .4.1 | Vital Signs | 8 |
| 9.2 | .4.2 | Laboratory Tests | 9 |
| 9.2 | .4.3 | Other Observations | 9 |
| 9.2 | 5 | Adverse Events (AEs) | 9 |
| 10.0 | An | alysis Items and Methods | 11 |
| 10.1 | Ma | atters on Patient Composition | 11 |
| 10.2 | | tient Demographics and Baseline Characteristics | |
| 10.3 | Tre | eatment Given | 11 |
| 10.4 | Ma | atters on Safety | 11 |
| 10. | 4.1 | Occurrence of Adverse Events | 11 |
| 10. | 4.2 | Factors that May Affect the Safety | 12 |
| 10.5 | Ma | atters on Efficacy | 12 |
| 10. | 5.1 | Office Blood Pressure | 12 |
| 10. | .5.2 | Factors that May Affect the Efficacy | |
| 11.0 | Pos | sting of Survey Information | 12 |
| 12.0 | Org | ganization | 12 |

| 12.1 | Administrative Manager | 12 |
|----------|------------------------------------------------|----|
| 12.2 | Central Registration Center | 12 |
| 13.0 | Contract Research Organizations | 12 |
| 14.0 | Other Necessary Matters | 13 |
| 14.1 | Revision of the Protocol | 13 |
| 14.2 | Actions to be Taken for Problems and Questions | 13 |
| Appendix | Observation schedule | |

#### 1.0 Background

Since drugs for hypertension are generally used for a long period of time, the safety of long-term use must be established. While the safety of long-term use of Zacras Combination Tablets LD & HD (hereinafter referred to as Zacras Combination Tablets) was already evaluated in a Japanese Phase III long-term clinical study (duration of treatment: 52 weeks, number of evaluated subjects: 368), it is necessary to evaluate the safety in more patients in clinical settings after marketing, a population that, unlike the study population, receive the drug in diverse situations.

Accordingly, a specified drug-use survey (hereinafter referred to as the survey) is planned to evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in hypertensive patients in daily medical practice. This survey will be conducted in compliance with Good Post-marketing Study Practice (GPSP) ordinance and related requirements.

#### 2.0 Objectives

To evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in hypertensive patients in daily medical practice

#### 3.0 Planned Sample Size and Rationale

#### 3.1 Planned Sample Size

1,000 patients

#### 3.2 Rationale

Patient populations identified as important missing information from Japanese clinical studies of Zacras Combination Tablets are patients with renal impairment, patients with hepatic impairment, and elderly patients ( $\geq 75$  years old). The sample size required to evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in these patient populations was calculated by reference to previous results. More specifically, according to final tabulation (number of patients included in safety evaluation: 3,300) in a previous specified drug-use survey (long-term use survey in hypertension) of a fixed-dose combination (UNISIA Combination Tablets) of an angiotensin receptor blocker (ARB) (candesartan) and a Ca antagonist (amlodipine), which belongs to the pharmacologically same class as Zacras Combination Tablets, patients with renal impairment, patients with hepatic impairment, and elderly patients (and those  $\geq$ 75 years old) accounted for 6.9%, 11.5%, and 65.2% (36.8%) of all patients, respectively. According to final tabulation (number of patients included in safety evaluation: 4,152) in a drug use-results survey of candesartan alone (BLOPRESS Tablets), patients with renal impairment, patients with hepatic impairment, and elderly patients (and those  $\geq 75$  years old) accounted for 9.5%, 10.6%, and 53.2% (22.1%), respectively. With a target sample size of 1,000 patients for the present survey, 70 patients with renal impairment, 100 patients with hepatic impairment, and 500 elderly patients (and 200 patients ≥75 years old)

are expected to be collected, probably allowing the safety and efficacy evaluation in these populations. This calculation is not based on statistical estimation.

#### 4.0 Survey Population

The survey population consists of hypertensive patients who do not meet any of the exclusion criteria listed in Section 4.1. Refer to the "Precautions for Indication" (presented below) and "Precautions" sections in the package insert.

<Pre><Precautions for Indication>

Zacras Combination Tablets should not be used as the first-line treatment of hypertension. An excessive drop in blood pressure may occur.

#### 4.1 Exclusion Criteria

Patients who meet any of the following criteria should be excluded from the survey:

- (1) Patients with a history of hypersensitivity to any of the ingredients of Zacras Combination Tablets or other dihydropyridines
- (2) Patients who are or may be pregnant
- (3) Diabetic patients taking aliskiren fumarate (excluding those with markedly poor blood pressure control despite other antihypertensive treatments)

#### 5.0 Dosage and Administration

For adults, one Zacras Combination Tablet (20 mg/2.5 mg or 20 mg/5 mg of azilsartan/amlodipine) will be administered orally once daily. Zacras Combination Tablets should not be used as the first-line treatment of hypertension. Refer to the "Precautions for Dosage and Administration" (presented below) and "Precautions" sections in the package insert.

<Precautions for Dosage and Administration>

(1) It should be determined whether Zacras Combination Tablets are indicated for each patient individually based on the following Dosage and Administration and Precautions for Dosage and Administration of azilsartan and amlodipine besilate, as well as other relevant information:

Azilsartan

Dosage and Administration

For adults, azilsartan 20 mg should usually be administered orally once daily. The dose may be increased or reduced as appropriate based on age and symptoms, with the maximum daily dose being 40 mg.

Precautions for Dosage and Administration

It should be carefully determined whether or not azilsartan is indicated while keeping the hypotensive effect of azilsartan in mind. Initiation of treatment at a low dose below 20 mg should also be considered

Amlodipine besilate

•Hypertension

Dosage and Administration

For adults, amlodipine 2.5 to 5 mg should usually be administered orally once daily. The dose may be increased or reduced as appropriate based on symptoms. In the case of insufficient response, the dose may be increased up to 10 mg given once daily.

(2) As a general rule, switching to Zacras Combination Tablets should be considered for patients receiving azilsartan 20 mg with amlodipine 2.5 to 5 mg or patients with poor blood pressure control despite treatment with either one of these treatments.

#### 6.0 Planned Number of Medical Institutions by Department

Internal medicine and other departments Approximately 250 medical institutions

#### 7.0 Methods

7.1 Observation Period

12 months

#### 7.2 Request to and Contract with the Study Site

Request and contract for participation in the survey will be made using a paper case report form (CRF). A representative of Takeda Pharmaceutical Company Limited (hereinafter referred to as Takeda's representative) will explain the objectives, contents, and methods of the survey to the investigator based on "Request for cooperation for specified drug-use survey," "Implementation outline," "Patient registration form (sample)," and "Case report form (sample)" to enter into a written contract with the study site and request the study site to conduct a survey within a specified period.

#### 7.3 Method of Patient Registration

Patients will be registered using the central registration system via fax. After the start of the contract with the study site, the investigator shall register each patient for whom Zacras Combination Tablets are prescribed by faxing a patient registration form containing patient registration information (refer to Section 9.1) to the central registration center (refer to Section 12.2) within 14 days after prescription of Zacras Combination Tablets (day of prescription designated as day 0 and day following the day of prescription designated as 1 day after prescription). No patient can be registered before Zacras Combination Tablets are actually prescribed. Patients determined by the central registration center to be ineligible for any reason cannot be registered. The investigator shall register a new patient using a new patient registration form supplied by Takeda's representative.

Takeda's representative will supply a CRF, which will be issued after the central registration

center decides to register the relevant patient, to the investigator.

#### 7.4 Completion and Submission of Case Report Form

For each of all registered patients, the investigator shall complete and submit a CRF to Takeda Pharmaceutical within approximately 1 month after the end of the observation period. Any failure to confirm the intake of Zacras Combination Tablets shall be specified (no further information is required).

For patients discontinued from treatment with Zacras Combination Tablets for any reason during the observation period, the investigator shall complete and submit a CRF to Takeda Pharmaceutical within approximately 1 month after the end of required observation. For any patient discontinued from treatment with Zacras Combination Tablets due to an adverse event, the investigator shall complete and submit a CRF to Takeda Pharmaceutical after monitoring the patient as long after discontinuation of treatment as possible until the adverse event is confirmed to have resolved or be resolving.

#### 7.5 Actions to be Taken in Case of Serious Adverse Events

The investigator shall immediately communicate any serious adverse event in the observation period to Takeda's representative. In addition, the investigator shall provide detailed information at the request of Takeda's representative.

#### 8.0 Planned Period

Survey period: From June 2014 to 31 January 2017

Patient enrollment period: From June 2014 to 31 January 2016<sup>Note)</sup>

Note) Patient registration (receipt of a patient registration form via fax) will not be accepted on 1 February 2016 onwards even if Zacras Combination Tablets are prescribed by 31 January 2016.

If the number of patients enrolled in the survey reaches the planned sample size before 31 January 2016, acceptance of registration will be terminated before the end of the patient enrollment period. If the patient enrollment period is shortened, the survey period will be changed accordingly.

#### 9.0 Survey Items

The investigator shall enter the items listed below into the patient registration form and the CRF. The survey schedule is presented in Appendix.

#### 9.1 Entries into the Patient Registration Form

#### 1) Survey items

Name of the medical institution, name of a physician who completes the patient registration form, date of prescription of Zacras Combination Tablets, patient identification number, patient initials, sex, date of birth, assessment based on the inclusion criteria, assessment

based on the exclusion criteria, presence or absence of breast-feeding (only females)

2) Time points of survey

At patient registration

#### 9.2 Entries into the Case Report Form

#### 9.2.1 Cover of the Case Report Form

Date of final entry into the CRF, name of a physician who completes the CRF

#### 9.2.2 Patient Demographics and Baseline Characteristics

#### 1) Survey items

Time of diagnosis of hypertension, diagnostic category (at the start of treatment with Zacras Combination Tablets), predisposition to hypersensitivity (presence or absence and details), concurrent illness (presence or absence and details), medical history (presence or absence and details), height, body weight, smoking history, drinking history, presence or absence of breast-feeding (at the start of treatment with Zacras Combination Tablets) [only females]

2) Time points of survey

At the start of treatment with Zacras Combination Tablets

#### 9.2.3 Treatment Given

#### 1) Survey items

Details on the use of Zacras Combination Tablets (daily dose, duration of treatment, and reason for discontinuation of treatment), details on the use of other antihypertensive \* (presence or absence, name of the drug, daily dose, and duration of treatment), details on the use of concomitant non-antihypertensive drug (presence or absence, name of the drug, and purpose of use)

#### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

\* Period from 2 months before the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment) for details on the use of other antihypertensive

#### 9.2.4 Tests/Observations

#### 9.2.4.1 Vital Signs

1) Tests/observations

Office blood pressure (systolic/diastolic), pulse rate

2) Time points of survey

Time points of measurement at the start of treatment with Zacras Combination Tablets and after 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 months of treatment (or discontinuation of

treatment)

#### 9.2.4.2 Laboratory Tests

#### 1) Test parameters

White blood cell count, platelet count, aspartate aminotransferase (AST), alanine aminotransferase (ALT),  $\gamma$ -glutamyl transpeptidase ( $\gamma$ -GTP), serum creatinine, blood urea nitrogen (BUN), serum potassium

#### 2) Time points of survey

Time points of test from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

#### 9.2.4.3 Other Observations

#### 1) Observations

Presence or absence of pregnancy in the observation period (only females)

If pregnancy is detected during the observation period, treatment with Zacras Combination

Tablets should be discontinued immediately, and Takeda's representative should be

informed. The investigator shall provide detailed information (including information up to
delivery such as premature delivery, wherever possible) using a pregnancy sheet at the
request of Takeda's representative.

#### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

#### 9.2.5 Adverse Events (AEs)

#### 1) Survey items

Presence or absence of AE (refer to Table 1), AE term, date of onset, seriousness and reason for seriousness (refer to Table 2), presence or absence of discontinuation of treatment with Zacras Combination Tablets, date of outcome assessment, outcome, causal relationship to Zacras Combination Tablets\* (refer to Table 3)

Patients with "not resolved" or "unknown" outcome or "unevaluable" causal relationship should be followed up wherever possible.

#### Note) Additional points to consider for AEs

Abnormal worsening of target disease, for instance, worsening beyond the expected natural course of the disease, will be handled as an AE, but expected worsening of target disease should not be handled as an AE.

#### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of

<sup>\*</sup> For the causal relationship to Zacras Combination Tablets, the rationale for "not related" and the reason for "unevaluable" shall be collected.

#### Table 1 Definition of adverse events

An AE is defined as any untoward medical occurrence in a clinical investigation subject administered a drug; it does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavorable or unintended sign (e.g., abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.

The following are also handled as AEs:

- •Symptoms and so forth that occur in infants breast-fed by their mothers under treatment with a drug
- •Symptoms and so forth that occur in children treated with a drug
- · Symptoms and so forth that occur as a result of occupational exposure to a drug
- · Symptoms and so forth that occur after administration of counterfeit medicines of our ethical drugs

#### Table 2 Criteria for assessing seriousness

An AE satisfying any of the following is assessed as serious:

- 1. Results in death (death)
- 2. Is life-threatening (risk of death)
- 3. Requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization/prolonged hospitalization)
- 4. Results in persistent or significant disability/incapacity (disability)
- 5. Leads to a congenital anomaly/birth defect (congenital anomaly)
- 6. Is an important medical event according to 1 to 5 described above, including AEs in Takeda Medically Significant AE List

#### Takeda Medically Significant AE List

Acute liver failure

| Takeda Medicany Significant AE List | |
|---|---|
| •Acute respiratory failure/acute respiratory distress | •Anaphylactic shock |
| syndrome (ARDS) | |
| •Torsade de pointes / ventricular fibrillation / ventricular | •Acute renal failure |
| tachycardia | |
| •Malignant hypertension | •Pulmonary hypertension |
| •Convulsive seizures (including convulsion and epilepsy) | •Pulmonary fibrosis (including interstitial |
| | pneumonia) |
| •Agranulocytosis | •Neuroleptic malignant syndrome / |
| | malignant hyperthermia |
| •Aplastic anemia | •Spontaneous abortion / stillbirth and fetal |
| | death |
| •Toxic epidermal necrolysis / oculomucocutaneous | •Confirmed or suspected transmission of |
| syndrome (Stevens-Johnson syndrome) | infectious agent by a medicinal product |
| •Hepatic necrosis | •Confirmed or suspected endotoxin shock |

Table 3 Criteria for assessing the relationship of each adverse event to Zacras Combination Tablets

| Assessment | Criteria for assessment |
|---|---|
| | An AE that follows a reasonable temporal sequence from |
| | administration of a drug (including the course after withdrawal of the |
| Deleted | drug), or for which possible involvement of the drug can be argued, |
| Related | although factors other than the drug, such as underlying diseases, |
| | concurrent illnesses, concomitant drugs, and concomitant treatments, |
| | may also be responsible |
| | An AE that does not follow a reasonable temporal sequence from |
| Not related | administration of a drug and/or that can reasonably be explained by |
| Not related | other factors, such as underlying diseases, concurrent illnesses, |
| | concomitant drugs, and concomitant treatments |
| | Information necessary for evaluation, including temporal sequence |
| TT 1 11 | from administration of a drug (including the course after withdrawal |
| Unevaluable | of the drug), underlying diseases, concurrent illnesses, concomitant |
| | drugs, and concomitant treatments, is not sufficient. |

#### 10.0 Analysis Items and Methods

#### 10.1 Matters on Patient Composition

The number of enrolled patients, number of patients from whom the CRF is collected, number of patients included in safety/efficacy analysis, number of patients excluded from analysis, and reason for exclusion will be tabulated.

#### 10.2 Patient Demographics and Baseline Characteristics

Patient demographics and baseline characteristics, including sex, age, duration of disease, predisposition to hypersensitivity, and concurrent illness, will be tabulated.

#### 10.3 Treatment Given

Details on the use of Zacras Combination Tablets, details on the use of other antihypertensive, and details on the use of concomitant non-antihypertensive drug will be tabulated.

#### 10.4 Matters on Safety

For the safety analysis set, data will be tabulated as described below. AEs will be coded according to the MedDRA/J and summarized using preferred term (PT) and system organ class (SOC).

#### 10.4.1 Occurrence of Adverse Events

For AEs reported during the observation period, the incidence will be tabulated by type, time

of onset, seriousness, and causal relationship to Zacras Combination Tablets.

#### 10.4.2 Factors that May Affect the Safety

For AEs reported during the observation period, the incidence will be tabulated by patient background factors (e.g., sex, age, presence or absence of concurrent renal impairment, presence or absence of concurrent hepatic impairment) and treatment given (e.g., details on the use of Zacras Combination Tablets, details on the use of concomitant drug).

#### 10.5 Matters on Efficacy

For the efficacy analysis set, data will be tabulated as described below.

#### 10.5.1 Office Blood Pressure

For office blood pressure, measured value, change (measured value at each post-baseline time point of measurement - measured value at the start of treatment with Zacras Combination Tablets), and percentage change [(measured value at each time point of measurement - measured value at the start of treatment with Zacras Combination Tablets) ÷ measured value at the start of treatment with Zacras Combination Tablets × 100] at each time point of test will be tabulated.

#### 10.5.2 Factors that May Affect the Efficacy

Office blood pressure will be tabulated by patient background factors (e.g., sex, age) and treatment given (e.g., details on the use of Zacras Combination Tablets, details on the use of other antihypertensive).

#### 11.0 Posting of Survey Information

Takeda Pharmaceutical Company Limited will post survey information on Clinical Trials.gov and an open website (JAPIC-CTI\*) before starting the survey.

# 12.0 Organization 12.1 Administrative Manager PPD Takeda Pharmaceutical Company Limited 12.2 Central Registration Center PPD

#### 13.0 Contract Research Organization

PPD

<sup>\*</sup> Japan Pharmaceutical Information Center-Clinical Trials Information



#### 14.0 Other Necessary Matters

#### 14.1 Revision of the Protocol

During the survey, attention will be paid to comprehend the status of progression of the survey, presence or absence of unexpected adverse drug reactions (ADRs)/serious ADRs (based on precautions), presence or absence of increased incidence of certain ADRs, and appropriateness of survey items, and this protocol will be reviewed and revised if necessary. If partial change to dosage and administration or indications is approved during the survey, the necessity of revising the protocol will be discussed if necessary, and the protocol will be revised as needed.

#### 14.2 Actions to be Taken for Problems and Questions

If any safety or efficacy problem is detected, data will be carefully examined to discuss measures.

#### Appendix Observation schedule

| Time point of survey | | Observation period | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time point of survey | | | | | J | J | J | J. | J | J | J | J | J. | J | J. | Jo |
| Survey item | | At patient registration | Start of treatment | After 1 month of treatment | After 2 months of treatment | After 3 months of treatment | After 4 months of treatment | After 5 months of treatment | After 6 months of treatment | After 7 months of treatment | After 8 months of treatment | After 9 months of treatment | After 10 months of treatment | After 11 months of treatment | After 12 months of treatment | At discontinuation of treatment |
| | Date of prescription of Zacras | 0 | | | | | | | | | | | | | | |
| | Combination Tablets | | | | | | | | | | | | | | | |
| tion | Patient identification number | 0 | | | | | | | | | | | | | | |
| stra | Patient initials | 0 | | | | | | | | | | | | | | |
| regi | Sex | 0 | | | | | | | | | | | | | | |
| Patient registration | Date of birth | 0 | | | | | | | | | | | | | | |
| Pat | Inclusion/exclusion criteria | 0 | | | | | | | | | | | | | | |
| | Presence or absence of | 0 | | | | | | | | | | | | | | |
| | breast-feeding (only females) | | | | | | | | | | | | | | | |
| tics | Time of diagnosis of | | 0 | | | | | | | | | | | | | |
| demographics and baseline characteristics | hypertension | | | | | | | | | | | | | | | |
| narac | Diagnostic category | | 0 | | | | | | | | | | | | | |
| ine cl | Predisposition to hypersensitivity | | 0 | | | | | | | | | | | | | |
| asel | Concurrent illness | | 0 | | | | | | | | | | | | | |
| and l | Medical history | | 0 | | | | | | | | | | | | | |
| hics | Height, body weight | | 0 | | | | | | | | | | | | | |
| ograp | Smoking history | | 0 | | | | | | | | | | | | | |
| demo | Drinking history | | 0 | | | | | | | | | | | | | |
| Patient | Presence or absence of | | 0 | | | | | | | | | | | | | |
| Ра | breast-feeding (only females) | | | | | | | | | | | | | | | |
| ı, etc. | Details on the use of Zacras Combination Tablets | | • • | | | | | | | | | | 0 | | | |
| Treatment given, etc. | Details on the use of other antihypertensive | | • • | | | | | | | | <b></b> | 0 | | | | |
| Treatm | Details on the use of concomitant non-antihypertensive drug | | <b>←</b> | | | | | | 0 | | | | | | <b></b> | 0 |
| etc. | Office blood pressure | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| ns, e | Pulse rate | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Tests/observations, | White blood cell count | | • | | 4 | · | • | <b></b> | 0 | | <b>4</b> | <b>4</b> | • | • | | 0 |
| serv | Platelet count | | <b>←</b> ○ ○ → | | | | | | | | | 0 | | | | |
| ts/ob | AST | | • | | | | | | 0 | | | | | | <b></b> | 0 |
| Tes | ALT | | <b>—</b> | | | | | | 0 | | | | | | <b></b> | 0 |
| لـــــــا | - | | L | | | | | | | | | | | | | |

| γ-GTP | <b>4</b> | 0 | <b>\</b> |
|---|---|---|---|
| Serum creatinine | | 0 | • 0 |
| BUN | <b>←</b> | o | • 0 |
| Serum potassium | <b>—</b> | o | <b>&gt;</b> 0 |
| Presence or absence of pregnancy (only females) | <b>-</b> | o — | • 0 |
| Adverse event | 4 | o | ▶ ○ |

o : Performed

← ∘ Performed throughout the period

## Protocol for Specified Drug-Use Survey Specified Drug-Use Survey ("Long-Term Use Survey") on Zacras Combination Tablets LD & HD

Version number 2nd version
Date of 15 May 2014

preparation

**Sponsor** Takeda Pharmaceutical Company Limited

#### Table of Contents

| 1.0 | | Background | | 4 |
|---|---|---|---|---|
| 2.0 | Objectives | | ectives | 2 |
| 3.0 | | Plan | ned Sample Size and Rationale | 2 |
| 3. | 1 | Plan | ned Sample Size | 2 |
| 3.2 | 2 | Rati | onale | 2 |
| 4.0 | | Surv | rey Population | 4 |
| 4. | 1 | Excl | usion Criteria | 4 |
| 5.0 | | Dosa | age and Administration | 4 |
| 6.0 | 6.0 Planned Number of Me | | ned Number of Medical Institutions by Department | ( |
| 7.0 | Methods | | hods | ( |
| 7. | .1 Observation Period | | ervation Period | ( |
| 7.2 | 7.2 Request to and Contract with the Study Site | | uest to and Contract with the Study Site | ( |
| 7.3 | 3 | Met | hod of Patient Registration | ( |
| 7.4 | .4 Completion and Submission of Case | | pletion and Submission of Case Report Form | |
| 7.5 | 5 | Acti | ons to be Taken in Case of Serious Adverse Events | |
| 8.0 | .0 Planned Period | | ned Period | |
| 9.0 | | | vey Items | |
| 9. | 1 | Entr | ies into the Patient Registration Form | |
| 9.2 | 2 | Entr | ies into the Case Report Form | 8 |
| | 9.2.1 | | Cover of the Case Report Form | 8 |
| | 9.2.2 | 2 | Patient Demographics and Baseline Characteristics | 8 |
| | 9.2.3 | 3 | Treatment Given | 8 |
| | 9.2.4 | ļ | Tests/Observations | 8 |
| | 9.2.4 | 1.1 | Vital Signs | 8 |
| | 9.2.4 | 1.2 | Laboratory Tests | 9 |
| | 9.2.4 | 1.3 | Other Observations. | 9 |
| | 9.2.5 | 5 | Adverse Events (AEs) | 9 |
| 10.0 | | Ana | lysis Items and Methods | 11 |
| 10 | 1.1 | Matt | ters on Patient Composition1 | 11 |
| 10 | .2 | Patie | ent Demographics and Baseline Characteristics | 11 |
| 10 | | | | |
| 10 | .4 | | | 1 |
| | 10.4 | .1 | Occurrence of Adverse Events | . 2 |
| | 10.4 | .2 | Factors that May Affect the Safety | . 2 |
| 10 | .5 | | ters on Efficacy | |
| | 10.5 | | Office Blood Pressure | |
| | 10.5 | .2 | Factors that May Affect the Efficacy | |
| 11.0 | | Posting of Survey Information | | |
| 12.0 | | | anization 1 | - |

| 12.1 | Administrative Manager | 12 |
|----------|------------------------------------------------|----|
| 12.2 | Central Registration Center | 12 |
| 13.0 | Contract Research Organization | 13 |
| 14.0 | Other Necessary Matters | 13 |
| 14.1 | Revision of the Protocol | 13 |
| 14.2 | Actions to be Taken for Problems and Questions | 13 |
| Appendix | x Observation schedule | |

#### 1.0 Background

Since drugs for hypertension are generally used for a long period of time, the safety of long-term use must be established. While the safety of long-term use of Zacras Combination Tablets LD & HD (hereinafter referred to as Zacras Combination Tablets) was already evaluated in a Japanese Phase III long-term clinical study (duration of treatment: 52 weeks, number of evaluated subjects: 368), it is necessary to evaluate the safety in more patients in clinical settings after marketing, a population that, unlike the study population, receive the drug in diverse situations.

Accordingly, a specified drug-use survey (hereinafter referred to as the survey) is planned to evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in hypertensive patients in daily medical practice. This survey will be conducted in compliance with Good Post-marketing Study Practice (GPSP) ordinance and related requirements.

#### 2.0 Objectives

To evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in hypertensive patients in daily medical practice

#### 3.0 Planned Sample Size and Rationale

#### 3.1 Planned Sample Size

1,000 patients

#### 3.2 Rationale

Patient populations identified as important missing information from Japanese clinical studies of Zacras Combination Tablets are patients with renal impairment, patients with hepatic impairment, and elderly patients ( $\geq 75$  years old). The sample size required to evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in these patient populations was calculated by reference to previous results. More specifically, according to final tabulation (number of patients included in safety evaluation: 3,300) in a previous specified drug-use survey (long-term use survey in hypertension) of a fixed-dose combination (UNISIA Combination Tablets) of an angiotensin receptor blocker (ARB) (candesartan) and a Ca antagonist (amlodipine), which belongs to the pharmacologically same class as Zacras Combination Tablets, patients with renal impairment, patients with hepatic impairment, and elderly patients (and those  $\geq$ 75 years old) accounted for 6.9%, 11.5%, and 65.2% (36.8%) of all patients, respectively. According to final tabulation (number of patients included in safety evaluation: 4,152) in a drug use-results survey of candesartan alone (BLOPRESS Tablets), patients with renal impairment, patients with hepatic impairment, and elderly patients (and those  $\geq 75$  years old) accounted for 9.5%, 10.6%, and 53.2% (22.1%), respectively. With a target sample size of 1,000 patients for the present survey, 70 patients with renal impairment, 100 patients with hepatic impairment, and 500 elderly patients (and 200 patients ≥75 years old)

are expected to be collected, probably allowing the safety and efficacy evaluation in these populations. This calculation is not based on statistical estimation.

#### 4.0 Survey Population

The survey population consists of hypertensive patients who do not meet any of the exclusion criteria listed in Section 4.1. Refer to the "Precautions for Indication" (presented below) and "Precautions" sections in the package insert.

<Pre><Precautions for Indication>

Zacras Combination Tablets should not be used as the first-line treatment of hypertension. An excessive drop in blood pressure may occur.

#### 4.1 Exclusion Criteria

Patients who meet any of the following criteria should be excluded from the survey:

- (1) Patients with a history of hypersensitivity to any of the ingredients of Zacras Combination Tablets or other dihydropyridines
- (2) Patients who are or may be pregnant
- (3) Diabetic patients taking aliskiren fumarate (excluding those with markedly poor blood pressure control despite other antihypertensive treatments)

#### 5.0 Dosage and Administration

For adults, one Zacras Combination Tablet (20 mg/2.5 mg or 20 mg/5 mg of azilsartan/amlodipine) will be administered orally once daily. Zacras Combination Tablets should not be used as the first-line treatment of hypertension. Refer to the "Precautions for Dosage and Administration" (presented below) and "Precautions" sections in the package insert.

<Precautions for Dosage and Administration>

(1) It should be determined whether Zacras Combination Tablets are indicated for each patient individually based on the following Dosage and Administration and Precautions for Dosage and Administration of azilsartan and amlodipine besilate, as well as other relevant information:

Azilsartan

Dosage and Administration

For adults, azilsartan 20 mg should usually be administered orally once daily. The dose may be increased or reduced as appropriate based on age and symptoms, with the maximum daily dose being 40 mg.

Precautions for Dosage and Administration

It should be carefully determined whether or not azilsartan is indicated while keeping the hypotensive effect of azilsartan in mind. Initiation of treatment at a low dose below 20 mg should also be considered.
Amlodipine besilate

•Hypertension

Dosage and Administration

For adults, amlodipine 2.5 to 5 mg should usually be administered orally once daily. The dose may be increased or reduced as appropriate based on symptoms. In the case of insufficient response, the dose may be increased up to 10 mg given once daily.

- (2) As a general rule, switching to Zacras Combination Tablets should be considered for patients receiving azilsartan 20 mg with amlodipine 2.5 to 5 mg or patients with poor blood pressure control despite treatment with either one of these treatments.
- 6.0 Planned Number of Medical Institutions by Department

Internal medicine and other departments Approximately 250 medical institutions

- 7.0 Methods
  - 7.1 Observation Period

12 months

### 7.2 Request to and Contract with the Study Site

Request and contract for participation in the survey will be made using a paper case report form (CRF). A medical representative of Takeda Pharmaceutical Company Limited (hereinafter referred to as Takeda's MR) will explain the objectives, contents, and methods of the survey to the investigator based on "Request for cooperation for specified drug-use survey," "Implementation outline," "Patient registration form (sample)," and "Case report form (sample)" to enter into a written contract with the study site and request the study site to conduct a survey within a specified period.

### 7.3 Method of Patient Registration

Patients will be registered using the central registration system via fax. After the start of the contract with the study site, the investigator shall register each patient for whom Zacras Combination Tablets are prescribed by faxing a patient registration form containing patient registration information (refer to Section 9.1) to the central registration center (refer to Section 12.2) within 14 days after prescription of Zacras Combination Tablets (day of prescription designated as day 0 and day following the day of prescription designated as 1 day after prescription). No patient can be registered before Zacras Combination Tablets are actually prescribed. Patients determined by the central registration center to be ineligible for any reason cannot be registered. The investigator shall register a new patient using a new patient registration form supplied by Takeda's MR.

Takeda's MR will supply a CRF, which will be issued after the central registration center

decides to register the relevant patient, to the investigator.

### 7.4 Completion and Submission of Case Report Form

For each of all registered patients, the investigator shall complete and submit a CRF to Takeda's MR within approximately 1 month after the end of the observation period. Any failure to confirm the intake of Zacras Combination Tablets shall be specified (no further information is required).

For patients discontinued from treatment with Zacras Combination Tablets for any reason during the observation period, the investigator shall complete and submit a CRF to Takeda's MR within approximately 1 month after the end of required observation. For any patient discontinued from treatment with Zacras Combination Tablets due to an adverse event, the investigator shall complete and submit a CRF to Takeda's MR after monitoring the patient as long after discontinuation of treatment as possible until the adverse event is confirmed to have resolved or be resolving.

### 7.5 Actions to be Taken in Case of Serious Adverse Events

The investigator shall immediately communicate any serious adverse event in the observation period to Takeda's MR. In addition, the investigator shall provide detailed information at the request of Takeda's MR.

### 8.0 Planned Period

Survey period: From June 2014 to 31 January 2017

Patient enrollment period: From June 2014 to 31 January 2016<sup>Note)</sup>

Note) Patient registration (receipt of a patient registration form via fax) will not be accepted on 1 February 2016 onwards even if Zacras Combination Tablets are prescribed by 31 January 2016.

If the number of patients enrolled in the survey reaches the planned sample size before 31 January 2016, acceptance of registration will be terminated before the end of the patient enrollment period. If the patient enrollment period is shortened, the survey period will be changed accordingly.

### 9.0 Survey Items

The investigator shall enter the items listed below into the patient registration form and the CRF. The survey schedule is presented in Appendix.

### 9.1 Entries into the Patient Registration Form

### 1) Survey items

Name of the medical institution, name of a physician who completes the patient registration form, date of prescription of Zacras Combination Tablets, patient identification number, patient initials, sex, date of birth, assessment based on the inclusion criteria, assessment

based on the exclusion criteria, presence or absence of breast-feeding (only females)

2) Time points of survey

At patient registration

### 9.2 Entries into the Case Report Form

### 9.2.1 Cover of the Case Report Form

Date of final entry into the CRF, name of a physician who completes the CRF

### 9.2.2 Patient Demographics and Baseline Characteristics

### 1) Survey items

Time of diagnosis of hypertension, diagnostic category (at the start of treatment with Zacras Combination Tablets), predisposition to hypersensitivity (presence or absence and details), concurrent illness (presence or absence and details), medical history (presence or absence and details), height, body weight, smoking history, drinking history, presence or absence of breast-feeding (at the start of treatment with Zacras Combination Tablets) [only females]

2) Time points of survey

At the start of treatment with Zacras Combination Tablets

### 9.2.3 Treatment Given

### 1) Survey items

Details on the use of Zacras Combination Tablets (daily dose, duration of treatment, and reason for discontinuation of treatment), details on the use of other antihypertensive \* (presence or absence, name of the drug, daily dose, and duration of treatment), details on the use of concomitant non-antihypertensive drug (presence or absence, name of the drug, and purpose of use)

### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

\* Period from 2 months before the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment) for details on the use of other antihypertensive

### 9.2.4 Tests/Observations

### 9.2.4.1 Vital Signs

1) Tests/observations

Office blood pressure (systolic/diastolic), pulse rate

2) Time points of survey

Time points of measurement at the start of treatment with Zacras Combination Tablets and after 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 months of treatment (or discontinuation of

treatment)

### 9.2.4.2 Laboratory Tests

### 1) Test parameters

White blood cell count, platelet count, aspartate aminotransferase (AST), alanine aminotransferase (ALT),  $\gamma$ -glutamyl transpeptidase ( $\gamma$ -GTP), serum creatinine, blood urea nitrogen (BUN), serum potassium

### 2) Time points of survey

Time points of test from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

### 9.2.4.3 Other Observations

### 1) Observations

Presence or absence of pregnancy in the observation period (only females)

If pregnancy is detected during the observation period, treatment with Zacras Combination Tablets should be discontinued immediately, and Takeda's MR should be informed. The investigator shall provide detailed information (including information up to delivery such as premature delivery, wherever possible) using a pregnancy sheet at the request of Takeda's MR.

### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

### 9.2.5 Adverse Events (AEs)

### 1) Survey items

Presence or absence of AE (refer to Table 1), AE term, date of onset, seriousness and reason for seriousness (refer to Table 2), presence or absence of discontinuation of treatment with Zacras Combination Tablets, date of outcome assessment, outcome, causal relationship to Zacras Combination Tablets\* (refer to Table 3)

Patients with "not resolved" or "unknown" outcome or "unevaluable" causal relationship should be followed up wherever possible.

### Note) Additional points to consider for AEs

Abnormal worsening of target disease, for instance, worsening beyond the expected natural course of the disease, will be handled as an AE, but expected worsening of target disease should not be handled as an AE.

### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of

<sup>\*</sup> For the causal relationship to Zacras Combination Tablets, the rationale for "not related" and the reason for "unevaluable" shall be collected.

### Table 1 Definition of adverse events

An AE is defined as any untoward medical occurrence in a clinical investigation subject administered a drug; it does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavorable or unintended sign (e.g., abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.

The following are also handled as AEs:

- •Symptoms and so forth that occur in infants breast-fed by their mothers under treatment with a drug
- •Symptoms and so forth that occur in children treated with a drug
- •Symptoms and so forth that occur as a result of occupational exposure to a drug
- •Symptoms and so forth that occur after administration of counterfeit medicines of our ethical drugs

### **Table 2 Criteria for assessing seriousness**

An AE satisfying any of the following is assessed as serious:

- 1. Results in death (death)
- 2. Is life-threatening (risk of death)
- 3. Requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization/prolonged hospitalization)
- 4. Results in persistent or significant disability/incapacity (disability)
- 5. Leads to a congenital anomaly/birth defect (congenital anomaly)
- 6. Is an important medical event according to 1 to 5 described above, including AEs in Takeda Medically Significant AE List

### Takeda Medically Significant AE List

Acute liver failure

| Takeua Medically Significant AE List | |
|---|---|
| •Acute respiratory failure/acute respiratory distress | •Anaphylactic shock |
| syndrome (ARDS) | |
| •Torsade de pointes / ventricular fibrillation / ventricular | •Acute renal failure |
| tachycardia | |
| •Malignant hypertension | •Pulmonary hypertension |
| •Convulsive seizures (including convulsion and epilepsy) | •Pulmonary fibrosis (including interstitial |
| | pneumonia) |
| •Agranulocytosis | •Neuroleptic malignant syndrome / |
| | malignant hyperthermia |
| •Aplastic anemia | •Spontaneous abortion / stillbirth and fetal |
| | death |
| •Toxic epidermal necrolysis / oculomucocutaneous | •Confirmed or suspected transmission of |
| syndrome (Stevens-Johnson syndrome) | infectious agent by a medicinal product |
| •Hepatic necrosis | •Confirmed or suspected endotoxin shock |

Table 3 Criteria for assessing the relationship of each adverse event to Zacras Combination Tablets

| Assessment | Criteria for assessment |
|---|---|
| | An AE that follows a reasonable temporal sequence from |
| | administration of a drug (including the course after withdrawal of the |
| Dalata d | drug), or for which possible involvement of the drug can be argued, |
| Related | although factors other than the drug, such as underlying diseases, |
| | concurrent illnesses, concomitant drugs, and concomitant treatments, |
| | may also be responsible |
| | An AE that does not follow a reasonable temporal sequence from |
| | administration of a drug and/or that can reasonably be explained by |
| Not related | other factors, such as underlying diseases, concurrent illnesses, |
| | concomitant drugs, and concomitant treatments |
| | Information necessary for evaluation, including temporal sequence |
| T. 1 11 | from administration of a drug (including the course after withdrawal |
| Unevaluable | of the drug), underlying diseases, concurrent illnesses, concomitant |
| | drugs, and concomitant treatments, is not sufficient. |

### 10.0 Analysis Items and Methods

### 10.1 Matters on Patient Composition

The number of enrolled patients, number of patients from whom the CRF is collected, number of patients included in safety/efficacy analysis, number of patients excluded from analysis, and reason for exclusion will be tabulated.

### 10.2 Patient Demographics and Baseline Characteristics

Patient demographics and baseline characteristics, including sex, age, duration of disease, predisposition to hypersensitivity, and concurrent illness, will be tabulated.

### 10.3 Treatment Given

Details on the use of Zacras Combination Tablets, details on the use of other antihypertensive, and details on the use of concomitant non-antihypertensive drug will be tabulated.

### 10.4 Matters on Safety

For the safety analysis set, data will be tabulated as described below. AEs will be coded according to the MedDRA/J and summarized using preferred term (PT) and system organ class (SOC).

### 10.4.1 Occurrence of Adverse Events

For AEs reported during the observation period, the incidence will be tabulated by type, time of onset, seriousness, and causal relationship to Zacras Combination Tablets.

### 10.4.2 Factors that May Affect the Safety

For AEs reported during the observation period, the incidence will be tabulated by patient background factors (e.g., sex, age, presence or absence of concurrent renal impairment, presence or absence of concurrent hepatic impairment) and treatment given (e.g., details on the use of Zacras Combination Tablets, details on the use of concomitant drug).

### 10.5 Matters on Efficacy

For the efficacy analysis set, data will be tabulated as described below.

### 10.5.1 Office Blood Pressure

For office blood pressure, measured value, change (measured value at each post-baseline time point of measurement - measured value at the start of treatment with Zacras Combination Tablets), and percentage change [(measured value at each time point of measurement - measured value at the start of treatment with Zacras Combination Tablets)  $\div$  measured value at the start of treatment with Zacras Combination Tablets  $\times$  100] at each time point of test will be tabulated.

### 10.5.2 Factors that May Affect the Efficacy

Office blood pressure will be tabulated by patient background factors (e.g., sex, age) and treatment given (e.g., details on the use of Zacras Combination Tablets, details on the use of other antihypertensive).

### 11.0 Posting of Survey Information

Takeda Pharmaceutical Company Limited will post survey information on Clinical Trials.gov and an open website (JAPIC-CTI\*) before starting the survey.

# 12.0 Organization

| 12.1<br>PPD | Administrative Manager | |
|-------------|-----------------------------|-----------------------|
| | | Takeda Pharmaceutical |
| Coı | mpany Limited | |
| 12.2<br>PPD | Central Registration Center | |
| 110 | | |

<sup>\*</sup> Japan Pharmaceutical Information Center-Clinical Trials Information

# 13.0 Contract Research Organization

### Other Necessary Matters 14.0

### 14.1 Revision of the Protocol

During the survey, attention will be paid to comprehend the status of progression of the survey, presence or absence of unexpected adverse drug reactions (ADRs)/serious ADRs (based on precautions), presence or absence of increased incidence of certain ADRs, and appropriateness of survey items, and this protocol will be reviewed and revised if necessary. If partial change to dosage and administration or indications is approved during the survey, the necessity of revising the protocol will be discussed if necessary, and the protocol will be revised as needed.

### 14.2 Actions to be Taken for Problems and Questions

If any safety or efficacy problem is detected, data will be carefully examined to discuss measures.

# Appendix Observation schedule

| | Time point of survey | | | | | | Ol | oserv | ation | perio | od | , | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Time point of survey | ion | t | | £ | f | Į. | f | f | f | f | f | JC | J( | JC | Jo |
| Sur | vey item | At patient registration | Start of treatment | After 1 month of treatment | After 2 months of treatment | After 3 months of treatment | After 4 months of treatment | After 5 months of treatment | After 6 months of treatment | After 7 months of treatment | After 8 months of treatment | After 9 months of treatment | After 10 months of treatment | After 11 months of treatment | After 12 months of treatment | At discontinuation of treatment |
| | Date of prescription of Zacras | 0 | | | | | | | | | | | | | | |
| | Combination Tablets | | | | | | | | | | | | | ļ | | |
| tion | Patient identification number | 0 | | | | | | | | | | | | | | |
| stra | Patient initials | 0 | | | | | | | | | | | | | | |
| regi | Sex | 0 | | | | | | | | | | | | | | |
| Patient registration | Date of birth | 0 | ļ | ļ | | ļ | ļ | ļ | | ļ | ļ | <u> </u> | <u> </u> | <u> </u> | <u> </u> | |
| Pati | Inclusion/exclusion criteria | 0 | | | | | | | | | | | | | | |
| | Presence or absence of | 0 | | | | | | | | | | | | | | |
| | breast-feeding (only females) | | | | | | | | | | | | | | | |
| ics | Time of diagnosis of | | 0 | | | | | | | | | | | | | |
| terist | hypertension | | | | | | | | | | | | | | | |
| aracı | Diagnostic category | | 0 | | | | | | | | | | | | | |
| ne ch | Predisposition to hypersensitivity | | 0 | | | | | | | | | | | | | |
| aseli | Concurrent illness | | 0 | | | | | | | | | | | | | |
| demographics and baseline characteristics | Medical history | | 0 | | | | | | | | | | | | | |
| nics a | Height, body weight | | 0 | | | | | | | | | | | | | |
| grapl | Smoking history | | 0 | | | | | | | | | | | | | |
| lemo | Drinking history | | 0 | | | | | | | | | | | | | |
| Patient o | Presence or absence of | | 0 | | | | | | | | | | | | | |
| Pati | breast-feeding (only females) | | | | | | | | | | | | | L | L | |
| n, etc. | Details on the use of Zacras Combination Tablets | | • | | | | | | 0 | | | | | _ | - | 0 |
| Treatment given, | Details on the use of other antihypertensive | | <b>-</b> | | | | | | 0 | | | | | | <b>&gt;</b> | 0 |
| Treatm | Details on the use of concomitant non-antihypertensive drug | | <b>-</b> | | | | | | 0 | | | | | | | 0 |
| ر.<br>د | Office blood pressure | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| ıs, etc. | Pulse rate | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Tests/observations, | White blood cell count | | <b>—</b> | 1 | 1 | I | 1 | L | 0 | <u> </u> | 1 | 1 | 1 | 1 | | 0 |
| serva | Platelet count | | <b>—</b> | | | | | | o | | | | | | | 0 |
| s/ops | AST | | <b>—</b> | | | | | | | | | | | | | 0 |
| Test | ALT | | • | | | | | | | | | | | | | 0 |
| | ALI | | | | | | | | 0 | | | | | | _ | |

| γ-GTP | <b> </b> | 0 | <b>→</b> |
|-------------------------------------------------|----------|---|-------------|
| Serum creatinine | <b> </b> | 0 | <b>&gt;</b> |
| BUN | <b>—</b> | o | • 0 |
| Serum potassium | <b>—</b> | o | • 0 |
| Presence or absence of pregnancy (only females) | <b>-</b> | 0 | |
| Adverse event | <b>-</b> | o | • ( |

o : Performed

← ○ → Performed throughout the period

# Protocol for Specified Drug-Use Survey Specified Drug-Use Survey ("Long-Term Use Survey") on Zacras Combination Tablets LD & HD

Version number 1st version
Date of 8 April 2014

preparation

**Sponsor** Takeda Pharmaceutical Company Limited

## Table of Contents

| 1.0 | | Bacl | kground | 4 |
|---|---|---|---|---|
| 2.0 | | Obje | ectives | 2 |
| 3.0 | | Plan | ned Sample Size and Rationale | 2 |
| 3.1 | 1 | Plan | ned Sample Size | 2 |
| 3.2 | 2 | Rati | onale | 2 |
| 4.0 | | Surv | rey Population | 4 |
| 4.1 | 1 | Excl | usion Criteria | 4 |
| 5.0 | | Dosa | age and Administration | 4 |
| 6.0 | | Plan | ned Number of Medical Institutions by Department | ( |
| 7.0 | | Met | hods | ( |
| 7.1 | 1 | Obs | ervation Period | ( |
| 7.2 | 2 | Req | uest to and Contract with the Study Site | ( |
| 7.3 | 3 | Met | hod of Patient Registration | ( |
| 7.4 | 4 | Con | pletion and Submission of Case Report Form | |
| 7.5 | 5 | Acti | ons to be Taken in Case of Serious Adverse Events | 7 |
| 8.0 | | Plan | ned Period | |
| 9.0 | | Surv | vey Items | |
| 9.1 | 1 | Entr | ies into the Patient Registration Form | |
| 9.2 | 2 | Entr | ies into the Case Report Form | 8 |
| | 9.2.1 | | Cover of the Case Report Form | 8 |
| | 9.2.2 | 2 | Patient Demographics and Baseline Characteristics | 8 |
| | 9.2.3 | 3 | Treatment Given | 8 |
| | 9.2.4 | ļ | Tests/Observations | 8 |
| | 9.2.4 | 1.1 | Vital Signs | 8 |
| | 9.2.4 | 1.2 | Laboratory Tests | 9 |
| | 9.2.4 | 1.3 | Other Observations | 9 |
| | 9.2.5 | 5 | Adverse Events (AEs) | 9 |
| 10.0 | | Ana | lysis Items and Methods | 11 |
| 10 | 1.1 | Matt | ters on Patient Composition1 | 11 |
| 10 | .2 | Patie | ent Demographics and Baseline Characteristics | 11 |
| 10 | | | tment Given1 | |
| 10 | .4 | Mat | ters on Safety | 1 |
| | 10.4 | .1 | Occurrence of Adverse Events | . 2 |
| | 10.4 | .2 | Factors that May Affect the Safety | . 2 |
| 10 | .5 | | ters on Efficacy | |
| | 10.5 | | Office Blood Pressure | |
| | 10.5 | .2 | Factors that May Affect the Efficacy | |
| 11.0 | | Post | ing of Survey Information | |
| 12.0 | | | anization 1 | , |

| 12.1 | Administrative Manager | 12 |
|----------|------------------------------------------------|----|
| 12.2 | Central Registration Center | 12 |
| 13.0 | Contract Research Organization | 13 |
| 14.0 | Other Necessary Matters | 13 |
| 14.1 | Revision of the Protocol | 13 |
| 14.2 | Actions to be Taken for Problems and Questions | 13 |
| Appendix | x Observation schedule | |

### 1.0 Background

Since drugs for hypertension are generally used for a long period of time, the safety of long-term use must be established. While the safety of long-term use of Zacras Combination Tablets LD & HD (hereinafter referred to as Zacras Combination Tablets) was already evaluated in a Japanese Phase III long-term clinical study (duration of treatment: 52 weeks, number of evaluated subjects: 368), it is necessary to evaluate the safety in more patients in clinical settings after marketing, a population that, unlike the study population, receive the drug in diverse situations.

Accordingly, a specified drug-use survey (hereinafter referred to as the survey) is planned to evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in hypertensive patients in daily medical practice. This survey will be conducted in compliance with Good Post-marketing Study Practice (GPSP) ordinance and related requirements.

### 2.0 Objectives

To evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in hypertensive patients in daily medical practice

### 3.0 Planned Sample Size and Rationale

### 3.1 Planned Sample Size

1,000 patients

### 3.2 Rationale

Patient populations identified as important missing information from Japanese clinical studies of Zacras Combination Tablets are patients with renal impairment, patients with hepatic impairment, and elderly patients ( $\geq 75$  years old). The sample size required to evaluate the safety and efficacy of long-term use of Zacras Combination Tablets in these patient populations was calculated by reference to previous results. More specifically, according to final tabulation (number of patients included in safety evaluation: 3,300) in a previous specified drug-use survey (long-term use survey in hypertension) of a fixed-dose combination (UNISIA Combination Tablets) of an angiotensin receptor blocker (ARB) (candesartan) and a Ca antagonist (amlodipine), which belongs to the pharmacologically same class as Zacras Combination Tablets, patients with renal impairment, patients with hepatic impairment, and elderly patients (and those  $\geq$ 75 years old) accounted for 6.9%, 11.5%, and 65.2% (36.8%) of all patients, respectively. According to final tabulation (number of patients included in safety evaluation: 4,152) in a drug use-results survey of candesartan alone (BLOPRESS Tablets), patients with renal impairment, patients with hepatic impairment, and elderly patients (and those  $\geq 75$  years old) accounted for 9.5%, 10.6%, and 53.2% (22.1%), respectively. With a target sample size of 1,000 patients for the present survey, 70 patients with renal impairment, 100 patients with hepatic impairment, and 500 elderly patients (and 200 patients ≥75 years old)

are expected to be collected, probably allowing the safety and efficacy evaluation in these populations. This calculation is not based on statistical estimation.

### 4.0 Survey Population

The survey population consists of hypertensive patients who do not meet any of the exclusion criteria listed in Section 4.1. Refer to the "Precautions for Indication" (presented below) and "Precautions" sections in the package insert.

<Pre><Precautions for Indication>

Zacras Combination Tablets should not be used as the first-line treatment of hypertension. An excessive drop in blood pressure may occur.

### 4.1 Exclusion Criteria

Patients who meet any of the following criteria should be excluded from the survey:

- (1) Patients with a history of hypersensitivity to any of the ingredients of Zacras Combination Tablets or other dihydropyridines
- (2) Patients who are or may be pregnant
- (3) Diabetic patients taking aliskiren fumarate (excluding those with markedly poor blood pressure control despite other antihypertensive treatments)

### 5.0 Dosage and Administration

For adults, one Zacras Combination Tablet (20 mg/2.5 mg or 20 mg/5 mg of azilsartan/amlodipine) will be administered orally once daily. Zacras Combination Tablets should not be used as the first-line treatment of hypertension. Refer to the "Precautions for Dosage and Administration" (presented below) and "Precautions" sections in the package insert.

<Pre><Pre>cautions for Dosage and Administration>

(1) It should be determined whether Zacras Combination Tablets are indicated for each patient individually based on the following Dosage and Administration and Precautions for Dosage and Administration of azilsartan and amlodipine besilate, as well as other relevant information:

Azilsartan

Dosage and Administration

For adults, azilsartan 20 mg should usually be administered orally once daily. The dose may be increased or reduced as appropriate based on age and symptoms, with the maximum daily dose being 40 mg.

Precautions for Dosage and Administration

It should be carefully determined whether or not azilsartan is indicated while keeping the hypotensive effect of azilsartan in mind. Initiation of treatment at a low dose below 20 mg should also be considered.

Amlodipine besilate

•Hypertension

Dosage and Administration

For adults, amlodipine 2.5 to 5 mg should usually be administered orally once daily. The dose may be increased or reduced as appropriate based on symptoms. In the case of insufficient response, the dose may be increased up to 10 mg given once daily.

- (2) As a general rule, switching to Zacras Combination Tablets should be considered for patients receiving azilsartan 20 mg with amlodipine 2.5 to 5 mg or patients with poor blood pressure control despite treatment with either one of these treatments.
- 6.0 Planned Number of Medical Institutions by Department

Internal medicine and other departments Approximately 250 medical institutions

- 7.0 Methods
  - 7.1 Observation Period

12 months

### 7.2 Request to and Contract with the Study Site

Request and contract for participation in the survey will be made using a paper case report form (CRF). A medical representative of Takeda Pharmaceutical Company Limited (hereinafter referred to as Takeda's MR) will explain the objectives, contents, and methods of the survey to the investigator based on "Request for cooperation for specified drug-use survey," "Implementation outline," "Patient registration form (sample)," and "Case report form (sample)" to enter into a written contract with the study site and request the study site to conduct a survey within a specified period.

### 7.3 Method of Patient Registration

Patients will be registered using the central registration system via fax. After the start of the contract with the study site, the investigator shall register each patient for whom Zacras Combination Tablets are prescribed by faxing a patient registration form containing patient registration information (refer to Section 9.1) to the central registration center (refer to Section 12.2) within 14 days after prescription of Zacras Combination Tablets (day of prescription designated as day 0 and day following the day of prescription designated as 1 day after prescription). No patient can be registered before Zacras Combination Tablets are actually prescribed. Patients determined by the central registration center to be ineligible for any reason cannot be registered. The investigator shall register a new patient using a new patient registration form supplied by Takeda's MR.

Takeda's MR will supply a CRF, which will be issued after the central registration center

decides to register the relevant patient, to the investigator.

### 7.4 Completion and Submission of Case Report Form

For each of all registered patients, the investigator shall complete and submit a CRF to Takeda's MR within approximately 1 month after the end of the observation period. Any failure to confirm the intake of Zacras Combination Tablets shall be specified (no further information is required).

For patients discontinued from treatment with Zacras Combination Tablets for any reason during the observation period, the investigator shall complete and submit a CRF to Takeda's MR within approximately 1 month after the end of required observation. For any patient discontinued from treatment with Zacras Combination Tablets due to an adverse event, the investigator shall complete and submit a CRF to Takeda's MR after monitoring the patient as long after discontinuation of treatment as possible until the adverse event is confirmed to have resolved or be resolving.

### 7.5 Actions to be Taken in Case of Serious Adverse Events

The investigator shall immediately communicate any serious adverse event in the observation period to Takeda's MR. In addition, the investigator shall provide detailed information at the request of Takeda's MR.

### 8.0 Planned Period

Survey period: From June 2014 to 31 January 2017

Patient enrollment period: From June 2014 to 31 January 2016<sup>Note)</sup>

Note) Patient registration (receipt of a patient registration form via fax) will not be accepted on 1 February 2016 onwards even if Zacras Combination Tablets are prescribed by 31 January 2016.

If the number of patients enrolled in the survey reaches the planned sample size before 31 January 2016, acceptance of registration will be terminated before the end of the patient enrollment period. If the patient enrollment period is shortened, the survey period will be changed accordingly.

### 9.0 Survey Items

The investigator shall enter the items listed below into the patient registration form and the CRF. The survey schedule is presented in Appendix.

### 9.1 Entries into the Patient Registration Form

### 1) Survey items

Name of the medical institution, name of a physician who completes the patient registration form, date of prescription of Zacras Combination Tablets, patient identification number, patient initials, sex, date of birth, assessment based on the inclusion criteria, assessment

based on the exclusion criteria, presence or absence of breast-feeding (only females)

2) Time points of survey

At patient registration

### 9.2 Entries into the Case Report Form

### 9.2.1 Cover of the Case Report Form

Date of final entry into the CRF, name of a physician who completes the CRF

### 9.2.2 Patient Demographics and Baseline Characteristics

### 1) Survey items

Time of diagnosis of hypertension, diagnostic category (at the start of treatment with Zacras Combination Tablets), predisposition to hypersensitivity (presence or absence and details), concurrent illness (presence or absence and details), medical history (presence or absence and details), height, body weight, smoking history, drinking history, presence or absence of breast-feeding (at the start of treatment with Zacras Combination Tablets) [only females]

2) Time points of survey

At the start of treatment with Zacras Combination Tablets

### 9.2.3 Treatment Given

### 1) Survey items

Details on the use of Zacras Combination Tablets (daily dose, duration of treatment, and reason for discontinuation of treatment), details on the use of other antihypertensive \* (presence or absence, name of the drug, daily dose, and duration of treatment), details on the use of concomitant non-antihypertensive drug (presence or absence, name of the drug, and purpose of use)

### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

\* Period from 2 months before the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment) for details on the use of other antihypertensive

### 9.2.4 Tests/Observations

### 9.2.4.1 Vital Signs

1) Tests/observations

Office blood pressure (systolic/diastolic), pulse rate

2) Time points of survey

Time points of measurement at the start of treatment with Zacras Combination Tablets and after 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 months of treatment (or discontinuation of

treatment)

### 9.2.4.2 Laboratory Tests

### 1) Test parameters

White blood cell count, platelet count, aspartate aminotransferase (AST), alanine aminotransferase (ALT),  $\gamma$ -glutamyl transpeptidase ( $\gamma$ -GTP), serum creatinine, blood urea nitrogen (BUN), serum potassium

### 2) Time points of survey

Time points of test from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

### 9.2.4.3 Other Observations

### 1) Observations

Presence or absence of pregnancy in the observation period (only females)

If pregnancy is detected during the observation period, treatment with Zacras Combination Tablets should be discontinued immediately, and Takeda's MR should be informed. The investigator shall provide detailed information (including information up to delivery such as premature delivery, wherever possible) using a pregnancy sheet at the request of Takeda's MR.

### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of treatment (or discontinuation of treatment)

### 9.2.5 Adverse Events (AEs)

### 1) Survey items

Presence or absence of AE (refer to Table 1), AE term, date of onset, seriousness and reason for seriousness (refer to Table 2), presence or absence of discontinuation of treatment with Zacras Combination Tablets, date of outcome assessment, outcome, causal relationship to Zacras Combination Tablets\* (refer to Table 3)

Patients with "not resolved" or "unknown" outcome or "unevaluable" causal relationship should be followed up wherever possible.

### Note) Additional points to consider for AEs

Abnormal worsening of target disease, for instance, worsening beyond the expected natural course of the disease, will be handled as an AE, but expected worsening of target disease should not be handled as an AE.

### 2) Time points of survey

Period from the start of treatment with Zacras Combination Tablets to 12 months of

<sup>\*</sup> For the causal relationship to Zacras Combination Tablets, the rationale for "not related" and the reason for "unevaluable" shall be collected.

### Table 1 Definition of adverse events

An AE is defined as any untoward medical occurrence in a clinical investigation subject administered a drug; it does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavorable or unintended sign (e.g., abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.

The following are also handled as AEs:

- •Symptoms and so forth that occur in infants breast-fed by their mothers under treatment with a drug
- •Symptoms and so forth that occur in children treated with a drug
- •Symptoms and so forth that occur as a result of occupational exposure to a drug
- •Symptoms and so forth that occur after administration of counterfeit medicines of our ethical drugs

### **Table 2 Criteria for assessing seriousness**

An AE satisfying any of the following is assessed as serious:

- 1. Results in death (death)
- 2. Is life-threatening (risk of death)
- 3. Requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization/prolonged hospitalization)
- 4. Results in persistent or significant disability/incapacity (disability)
- 5. Leads to a congenital anomaly/birth defect (congenital anomaly)
- 6. Is an important medical event according to 1 to 5 described above, including AEs in Takeda Medically Significant AE List

### Takeda Medically Significant AE List

Acute liver failure

| Takeda Medicany Significant AE List | |
|---|---|
| •Acute respiratory failure/acute respiratory distress | •Anaphylactic shock |
| syndrome (ARDS) | |
| •Torsade de pointes / ventricular fibrillation / ventricular | •Acute renal failure |
| tachycardia | |
| •Malignant hypertension | •Pulmonary hypertension |
| •Convulsive seizures (including convulsion and epilepsy) | •Pulmonary fibrosis (including interstitial |
| | pneumonia) |
| •Agranulocytosis | •Neuroleptic malignant syndrome / |
| | malignant hyperthermia |
| •Aplastic anemia | •Spontaneous abortion / stillbirth and fetal |
| | death |
| •Toxic epidermal necrolysis / oculomucocutaneous | •Confirmed or suspected transmission of |
| syndrome (Stevens-Johnson syndrome) | infectious agent by a medicinal product |
| •Hepatic necrosis | •Confirmed or suspected endotoxin shock |

Table 3 Criteria for assessing the relationship of each adverse event to Zacras Combination Tablets

| Assessment | Criteria for assessment |
|---|---|
| | An AE that follows a reasonable temporal sequence from |
| | administration of a drug (including the course after withdrawal of the |
| Dalata d | drug), or for which possible involvement of the drug can be argued, |
| Related | although factors other than the drug, such as underlying diseases, |
| | concurrent illnesses, concomitant drugs, and concomitant treatments, |
| | may also be responsible |
| | An AE that does not follow a reasonable temporal sequence from |
| | administration of a drug and/or that can reasonably be explained by |
| Not related | other factors, such as underlying diseases, concurrent illnesses, |
| | concomitant drugs, and concomitant treatments |
| | Information necessary for evaluation, including temporal sequence |
| T. 1 11 | from administration of a drug (including the course after withdrawal |
| Unevaluable | of the drug), underlying diseases, concurrent illnesses, concomitant |
| | drugs, and concomitant treatments, is not sufficient. |

### 10.0 Analysis Items and Methods

### 10.1 Matters on Patient Composition

The number of enrolled patients, number of patients from whom the CRF is collected, number of patients included in safety/efficacy analysis, number of patients excluded from analysis, and reason for exclusion will be tabulated.

### 10.2 Patient Demographics and Baseline Characteristics

Patient demographics and baseline characteristics, including sex, age, duration of disease, predisposition to hypersensitivity, and concurrent illness, will be tabulated.

### 10.3 Treatment Given

Details on the use of Zacras Combination Tablets, details on the use of other antihypertensive, and details on the use of concomitant non-antihypertensive drug will be tabulated.

### 10.4 Matters on Safety

For the safety analysis set, data will be tabulated as described below. AEs will be coded according to the MedDRA/J and summarized using preferred term (PT) and system organ class (SOC).

### 10.4.1 Occurrence of Adverse Events

For AEs reported during the observation period, the incidence will be tabulated by type, time of onset, seriousness, and causal relationship to Zacras Combination Tablets.

### 10.4.2 Factors that May Affect the Safety

For AEs reported during the observation period, the incidence will be tabulated by patient background factors (e.g., sex, age, presence or absence of concurrent renal impairment, presence or absence of concurrent hepatic impairment) and treatment given (e.g., details on the use of Zacras Combination Tablets, details on the use of concomitant drug).

### 10.5 Matters on Efficacy

For the efficacy analysis set, data will be tabulated as described below.

### 10.5.1 Office Blood Pressure

For office blood pressure, measured value, change (measured value at each post-baseline time point of measurement - measured value at the start of treatment with Zacras Combination Tablets), and percentage change [(measured value at each time point of measurement - measured value at the start of treatment with Zacras Combination Tablets)  $\div$  measured value at the start of treatment with Zacras Combination Tablets  $\times$  100] at each time point of test will be tabulated.

### 10.5.2 Factors that May Affect the Efficacy

Office blood pressure will be tabulated by patient background factors (e.g., sex, age) and treatment given (e.g., details on the use of Zacras Combination Tablets, details on the use of other antihypertensive).

### 11.0 Posting of Survey Information

Takeda Pharmaceutical Company Limited will post survey information on Clinical Trials.gov and an open website (JAPIC-CTI\*) before starting the survey.

### 12.0 Organization

| .o organization | |
|-----------------------------|-----------------------|
| 12.1 Administrative Manager | |
| PPD | |
| | Takeda Pharmaceutical |
| Company Limited | |
| 122 G 1 D | |

# 12.2 Central Registration Center

<sup>\*</sup> Japan Pharmaceutical Information Center-Clinical Trials Information

### 13.0 Contract Research Organization

PPI

### 14.0 Other Necessary Matters

### 14.1 Revision of the Protocol

During the survey, attention will be paid to comprehend the status of progression of the survey, presence or absence of unexpected adverse drug reactions (ADRs)/serious ADRs (based on precautions), presence or absence of increased incidence of certain ADRs, and appropriateness of survey items, and this protocol will be reviewed and revised if necessary. If partial change to dosage and administration or indications is approved during the survey, the necessity of revising the protocol will be discussed if necessary, and the protocol will be revised as needed.

### 14.2 Actions to be Taken for Problems and Questions

If any safety or efficacy problem is detected, data will be carefully examined to discuss measures.

# Appendix Observation schedule

| | Time point of survey | | | | | | Ol | oserv | ation | perio | od | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Time point of survey | nc<br>_ | | | _ | , | , | | | | | | J | J | J | Jc |
| Sur | vey item | At patient registration | Start of treatment | After 1 month of treatment | After 2 months of treatment | After 3 months of treatment | After 4 months of treatment | After 5 months of treatment | After 6 months of treatment | After 7 months of treatment | After 8 months of treatment | After 9 months of treatment | After 10 months of treatment | After 11 months of treatment | After 12 months of treatment | At discontinuation of treatment |
| | Date of prescription of Zacras | | | | | | | | | | | | | | | |
| | Combination Tablets | 0 | | | | | | | | | | | | | | |
| ion | Patient identification number | 0 | | | | | | | | | | | | | | |
| strat | Patient initials | 0 | | | | | | | | | | | | | | |
| regi | Sex | 0 | | | | | | | | | | | | | | |
| Patient registration | Date of birth | 0 | | | | | | | | | | | | | | |
| Pati | Inclusion/exclusion criteria | 0 | | | | | | | | | | | | | | |
| | Presence or absence of | 0 | | | | | | | | | | | | | | |
| | breast-feeding (only females) | | | | | L | | | | | | | | | _ | |
| tics | Time of diagnosis of | | 0 | | | | | | | | | | | | | |
| teris | hypertension | | | | | | | | | | | | | | | |
| arac | Diagnostic category | | 0 | | | | | | | | | | | | | |
| ıe ch | Predisposition to hypersensitivity | | 0 | | | | | | | | | | | | | |
| aselir | Concurrent illness | | 0 | | | | | | | | | | | | | |
| demographics and baseline characteristics | Medical history | | 0 | | | | | | | | | | | | | |
| ics a | Height, body weight | | 0 | | | | | | | | | | | | | |
| graph | Smoking history | | 0 | | | | | | | | | | | | | |
| emos | Drinking history | | 0 | | | | | | | | | | | | | |
| | Presence or absence of | | 0 | | | | | | | | | | | | | |
| Patient | breast-feeding (only females) | | | | | | | | | | | | | | | |
| n, etc. | Details on the use of Zacras Combination Tablets | | <b>←</b> | | | | | | 0 | | | | | | <b></b> | 0 |
| Treatment given, | Details on the use of other antihypertensive | | • | | | | | | 0 | | | | | | <b></b> | 0 |
| Treatm | Details on the use of concomitant non-antihypertensive drug | | • | | | | | | 0 | | | | | | | 0 |
| | Office blood pressure | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| ıs, etc. | Pulse rate | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Tests/observations, | White blood cell count | | <b>—</b> | 1 | 1 | L | I | L | 0 | · | 1 | 1 | 1 | 1 | | 0 |
| serv | Platelet count | | <b>—</b> | | | | | | o | | | | | | | 0 |
| qo/s | AST | | <b>—</b> | | | | | | | | | | | | | 0 |
| Test | ALT | | <b>——</b> | | | | | | | | | | | | <b>-</b> | . 0 |
| | ALI | | <u> </u> | | | | | | <u>U</u> | | | | | | | |

| γ-GTP | <b> </b> | 0 | • • |
|-------------------------------------------------|----------|---|-----|
| Serum creatinine | <b>—</b> | 0 | • 0 |
| BUN | <b>—</b> | o | • 0 |
| Serum potassium | <b>—</b> | o | • 0 |
| Presence or absence of pregnancy (only females) | <b>-</b> | 0 | • |
| Adverse event | <b>←</b> | o | • 0 |

o : Performed

← ∘ Performed throughout the period